CLINICAL TRIAL: NCT02843048
Title: BaSEIB Clinical Trial - Bariatric Surgery and Exercise Intervention Bone Trial
Brief Title: Bariatric Surgery and Exercise Bone Trial
Acronym: BaSEIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Hélder Fonseca, PhD, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PTDC/DTP-DES/0968/2014; POCI-01-0145-FEDER-016707 (Other Grant/Funding Number: FEDER/COMPETE)
Record Dates: First submitted 2016-07-14; First posted 2016-07-25 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Metabolic Bone Disease; Accidental Falls
Keywords: Osteoporosis; Bariatric Surgery; Physical exercise; Obesity
MeSH Terms: conditions — Obesity; Bone Diseases, Metabolic; Osteoporosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): Exercise training plus standard medical follow-up care
  Interventions: Behavioral: Exercise training program
- Standard medical care (Active Comparator): Standard medical follow-up care only
  Interventions: Behavioral: Standard medical care

INTERVENTIONS:
Behavioral: Exercise training program — Participants allocated to the "Exercise training plus standard medical care" group will undergo an exercise-training program of 11 months duration, 3 sessions/week, and 60 minutes/session, starting one month after the surgery. Each exercise session will be supervised and will include 5 major components: i) warm-up, ii) multidirectional jumps, iii) balance, iv) strength and, v) cool down. This structure is planned to meet two main objectives: i) enhance bone formation and, ii) reduce fall risk by improving muscle strength, cardiorespiratory fitness and balance.
  Arms: Exercise training
Behavioral: Standard medical care — Standard follow-up medical care following bariatric surgery
  Arms: Standard medical care

SUMMARY:
Despite being effective in weight reduction in severely obese patients, bariatric surgery (BS) negatively influences bone metabolism and increases the risk of falls thereby potentially increasing the risk of fracture. The mechanisms of BS induced bone loss are unknown but may be related to calcium and vitamin D malabsorption, changes in the energy regulation metabolism and gastrointestinal hormonal physiology. Since the etiology of BS induced bone loss is largely unknown, treatment relies mostly on calcium and vitamin D supplementation, which provide little benefit.

Exercise is an effective strategy to prevent bone mass losses in several health conditions. However, no study so far has examined the effects of an exercise-training program in the prevention of BS induced bone loss. The investigators main goal is to investigate the effects on bone metabolism and fracture risk of an exercise-training program specifically tailored to improve bone health and balance of patients that underwent BS. The investigators will perform a randomized controlled trial on obese patients (n=80; BMI>40 Kg.m-2) elected to BS. Patients will be randomly assigned into 2 groups i) a group receiving standard follow-up and medical care, or ii) a group that will undergo a 11 months' Exercise Training program designed to improve bone health and reduce fall risk plus the standard follow-up and medical care. All patients will be assessed i) before the surgery, ii) one month, iii) 6 months, and iv) 12 months after the surgery. Assessments include: biochemical markers of bone turnover (BTM), BMD, bone tissue biomechanical properties, hormones involved in the regulation of energy, gastrointestinal and bone metabolism, body composition, BMI, nutritional intake, balance, muscle strength, cardiorespiratory fitness and daily physical activity. These evaluations will allow the investigators to understand the effects of an exercise-training program on bone metabolism of BS patients, contributing also to further elucidate the mechanisms underlying BS induced bone loss and fracture risk increase. The investigators will use established methods in the literature as well as novel procedures, which will enable them to overcome some of the limitations of previous studies. At the end of the study the investigators expect to have collected consistent data about whether an exercise-training program is or is not able to effectively prevent BS induced bone losses and fracture risk increases.

DETAILED DESCRIPTION:
The investigators main goal is to determine if an Exercise-Training Intervention program (ETI) tailored to improve bone health, strength and balance, is effective in preventing Roux-en-Y gastric bypass (RYGB) induced fracture risk. To achieve this the investigators will perform a randomized clinical trial (RCT) on volunteer obese patients (BMI>35 Kg.m-2) undergoing RYGB that will be followed for 13-months (Figure 1). The patients will be recruited, operated and will receive follow-up medical care in the Department of General Surgery from the Centro Hospitalar de São João E.P.E (DSHSJ). After being elected for RYGB and if inclusion and exclusion criteria are met, patients who decide to join the study will be randomly assigned to either i) participate in a 11 months duration ETI tailored to improve bone health and reduce fall risk in addition to the standard follow-up medical care (MFU) (ETI+MFU group), or ii) will receive only MFU (control group). Recruiting patients from only one institution will increase the likelihood of all patients receiving the same surgical and MFU care, reducing the bias related to the use of different clinical protocols. The option to include only RYGB is also to reduce the bias associated with the surgical technique. Participants allocated to the ETI+MFU group will undergo an exercise-training program of 11 months duration, 3 sessions/week, and 60 minutes/session, starting one month after the surgery. Each exercise session will be supervised and will include 5 major components: i) warm-up, ii) multidirectional jumps, iii) balance, iv) strength and, v) cool down. This structure is planned to meet two main objectives: i) enhance bone formation and, ii) reduce fall risk by improving muscle strength, cardiorespiratory fitness and balance. The ETI will last almost 1 year because the effects of BS on bone metabolism have been shown to be greatest during the first postoperative year (1). As the investigators main objective is to understand, in a broad perspective, the possible therapeutic benefits that an ETI has on the BS patient bone health and fracture risk, the plan is to investigate several variables in this study (bone turnover markers, bone mineral content (BMC) and density (BMD), body composition, body mass index (BMI), nutritional intake, static balance, dynamic balance, muscle strength of the lower limbs and trunk, daily physical activity, cardiorespiratory fitness, bone derived hormones, hormones involved in phosphate and calcium metabolism, adipokines, gastrointestinal and energy-metabolism hormones and gonadal hormones). These will enable the investigators to comprehensively understand the metabolic changes following BS that might affect bone health, and how can exercise influence those changes potentially preventing fracture risk increases.

Each patient will be assessed 4 times during the study (Figure 1). Each assay will match the monitoring protocols already scheduled by the DSHSJ for all patients undergoing BS. The 1st evaluation will occur prior to BS, to gather pre-surgical state. The 2nd, 3rd and 4th evaluations will occur in the 1st (before the beginning of the exercise-training program for the patients allocated to the exercise intervention group), 6th and 12th months after bariatric surgery, respectively. The variables analyzed at each time point fit into four major categories: i) bone quality surrogates (BTM, BMD, bone biomechanical properties); ii) anthropometry (weight, height, body composition, nutritional intake; iii) fall risk (static and dynamic balance, muscle strength, cardiorespiratory fitness, daily physical activity), iv) hormones involved in calcium, bone and gastro-intestinal metabolism. Biochemical analysis will be performed in blood samples collected during follow up hospital visits. Biochemical markers of bone turnover (BTM) reflect the degree of bone remodeling and the balance between formation and resorption and are therefore surrogates of fracture risk. As BS profoundly affects body composition, gastrointestinal and energy-regulation physiology, and because adipose tissue and gut-associated hormones also influence bone metabolism, the investigators will determine how these hormones are affected by RYGB and exercise. By monitoring these variables the investigators will gain insight on the etiological mechanisms associated with BS induced bone loss and the therapeutic effects of exercise. BS also leads to a reduction in calcium and vitamin D absorption, which may result in increased bone resorption. The investigators will therefore also monitor Vitamin D, Parathyroid Hormone (PTH), calcium and phosphorous concentrations to determine how they are influenced by the ETI. Despite mechanical unloading due to the weight loss may contribute to bone loss following BS, there is no data supporting this mechanism. To investigate this relation, the investigators will also monitor serum sclerostin, a protein released by osteocytes in response to mechanical unloading that negatively regulates bone formation. To determine the effects of BS and exercise on skeletal muscle and adipose tissue mass, the investigators will measure body composition and BMI in all patients. As one of the investigators main goal is to investigate the effects of the ETI on fall risk, they also plan to determine the cardiorespiratory fitness and muscle strength in these patients since these variables have been previously shown to influence fall risk. Daily physical activity and nutritional intake will also be determined by accelerometer and food diary, respectively, in order to control for confounding variables. Despite the several caveats associated with the determination of BMD by DXA, the investigators plan to analyze this variable, as it will provide data that will enable them to compare their results with the results from previous studies. Nevertheless, the investigators plan to complement this information with the direct assessment of bone biomechanical properties, which until recently was only available in in vitro studies due to the invasive nature of the procedure. Bone micro-indentation is a newer technique that allows measuring bone tissue mechanical properties in the clinical setting, which reflects with higher accuracy the bone resistance to fracture (6). One of the main outcomes in this research is to investigate the effects of BS on fall risk, as there is almost no data on this issue. This will be accomplished by direct determination of static and dynamic balance by means of using a forces platform. By analyzing this broad set of parameters the investigators plan to contribute with a more thorough understanding of the effects of BS on bone metabolism and, most importantly, how can an exercise training program, specifically tailored to improve bone health and balance, can reduce the risk of bone fractures in these patients. Only by analyzing this broad number of parameters will the investigators be able to control the several confounding variables and gain deeper insight into the effects of BS and exercise on the bone metabolism of these patients, thereby contributing with a potently useful strategy for the management of skeletal health in BS patients.

ELIGIBILITY:
Inclusion Criteria:

* meet the referral criteria for bariatric surgery;
* BMI >40 kg.m-2 or >35 kg.m-2 with obesity-related comorbidities;
* Motivation to participate in the study, regardless to the allocation group

Exclusion Criteria:

* use of drugs that interfere with bone metabolism (i.e. bisphosphonates, teriparatide, calcitonin, hormone replacement therapy, chronic use of corticosteroids, thiazide diuretics);
* Unable to perform exercise of moderate intensity;
* Health condition that could be aggravated by exercise (i.e. uncontrolled arterial hypertension, severe kidney disease, class III New York Heart Association heart failure);
* Peri-menopausal status with last menstruation <1 year;
* Known metabolic bone disease (i.e. Osteogenesis Imperfecta, Paget bone disease);
* Concurrent participation in a structured exercise program (>30 min in duration >1 day/week);
* Pregnancy or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 12 months
  Assayed by dual energy x-ray absorptiometry (DXA); g/cm2
Biochemical marker of bone resorption | 12 months
  Collagen type 1 cross-linked C-telopeptide (CTX; ng/mL)
Bone Material Strength index (BMSi) | 12 months
  Normalized parameter of bone material's resistance to indentation (OsteoProbe RUO)

CONTACTS AND LOCATIONS:
Overall Officials: Hélder Fonseca, PhD, Principal Investigator — CIAFEL
Locations (1):
- Faculdade de Desporto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boppre G, Diniz-Sousa F, Veras L, Bezerra A, Devezas V, Preto J, Santos-Sousa H, Oliveira J, Fonseca H. Impact of a Multicomponent Exercise Training Program on Muscle Strength After Bariatric Surgery: A Randomized Controlled Trial. Obes Surg. 2024 May;34(5):1704-1716. doi: 10.1007/s11695-024-07173-w. Epub 2024 Mar 27. PMID 38532144
- See also: Project home page — https://ciafel.fade.up.pt/p_baseib.php